CLINICAL TRIAL: NCT02301533
Title: Provider and Peer Support Intervention to Improve ART Adherence Among Kenyan Men Who Have Sex With Men
Acronym: Shikamana
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Kenya Medical Research Institute (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Susan Graham, Associate Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 44022; 1R34MH099946 (NIH)
Record Dates: First submitted 2014-11-13; First posted 2014-11-26 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Medication Adherence
Keywords: HIV infection; antiretroviral therapy; adherence; men who have sex with men
MeSH Terms: conditions — Medication Adherence; HIV Infections; Homosexuality | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Shikamana Intervention (Experimental): The Shikamana Intervention consists of provider support (modified Next Step Counseling) and peer support (trained peer navigator) to promote adherence to antiretroviral therapy
  Interventions: Behavioral: Shikamana Intervention
- Standard Care (Other): The standard care arm will receive adherence counseling per standard Kenyan Ministry of Health guidelines, along with the recommendation to disclose to a family member or friend in order to obtain support
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Shikamana Intervention — See arm description
  Arms: Shikamana Intervention
Behavioral: Standard Care — See arm description
  Arms: Standard Care

SUMMARY:
Antiretroviral therapy (ART) can improve health, prevent complications due to HIV infection, and prevent HIV transmission by making people less infectious. Men who have sex with men (MSM) are at high risk for transmitting HIV, but face stigma and discrimination that can make ART adherence difficult. Our goal is to find out if an intervention involving provider counselling and support from an MSM peer will improve ART adherence and engagement in care among Kenyan MSM. This study will be carried out in the KEMRI clinic in Mtwapa with 70 MSM patient participants who reside in this area, identified through our outreach and testing programs in Mtwapa. Six providers and five peers who are trained for the intervention will also be consented in order to collect data on their feedback and help monitor the study. Our intervention consists of support from a trained peer with experience taking ART and enhanced counselling from providers that is aimed to motivate patients to improve and maintain their health. In an initial pilot test, we will implement our intervention with 10 MSM starting ART for the first time. After any needed revisions to research procedures and training, we will next conduct a small randomized controlled trial with 60 MSM patient participants to determine feasibility, acceptability, tolerability, and safety, and estimate an initial effect size for the adherence intervention. The 60 patient participants will be randomized to our intervention or to standard counselling care, and will be followed for 6 months to evaluate their ART adherence and retention in care. Providers and peers will give feedback at regular project meetings and in in-depth interviews after the pilot test and after the RCT. The work proposed for this project will be carried out over 2 years, from June 1, 2014 through May 31, 2016.

DETAILED DESCRIPTION:
Although men who have sex with men (MSM) are at very high risk for HIV globally, this group has only recently become an important focus of national HIV/AIDS programs in sub-Saharan Africa. While it is clear that antiretroviral therapy (ART) can reduce AIDS-related morbidity and mortality and prevent sexual transmission from HIV-infected MSM, this group faces significant stigma that can impede engagement in care. Based on qualitative research conducted in 2013-2014 in coastal Kenya, we have developed an intervention called "Shikamana" (a Kiswahili word meaning "to form a bond or stick together") to improve HIV treatment engagement, ART adherence, and clinical outcomes in this group. We now propose a 2-year study to pilot test and conduct an initial evaluation of this intervention. Our specific aims are to: 1) pilot test our evidence-based intervention for MSM and ensure that the intervention is feasible and acceptable to patient, peer, and provider participants; and 2) implement a small randomized controlled trial (RCT) of the resulting multi-component intervention versus standard care with 60 MSM patient participants. Ten patient participants will be followed in the pilot test for 3 months each, with monthly measurement of ART adherence, baseline and month 3 measurement of adherence correlates, and feedback from participants and staff on the intervention procedures. After fine-tuning of the intervention based on the pilot test, we will follow 60 MSM patient participants for 6 months each, with monthly measurement of ART adherence, baseline and quarterly measurement of adherence correlates, viral load testing at month 3 and month 6 as a biomarker of treatment success, and feedback from participants and staff on the intervention procedures. Findings from this formative 2-year study will provide qualitative data on the feasibility, acceptability, tolerability, safety, and quantitative data on preliminary effect sizes to test this intervention and its components in a fully powered RCT including a larger, more diverse sample of MSM from multiple sites in sub-Saharan Africa.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18 years or older
* Live or work in or around Mtwapa
* Kenyan nationality
* Engaged in any sex (manual, oral, anal) with a man during the past 12 months
* Documented HIV-1-infection
* Eligible for ART by current Kenyan guidelines
* Able to communicate in Swahili or English
* Willing to undergo randomization and participate in study procedures as outlined in the consent
* Not planning to move from area during the next 12 months To enhance study feasibility, we will recruit up to 30 men with prior ART experience. We will collect data on the duration of ART at the time of study enrolment.

Exclusion Criteria:

* Inability to understand the research, as assessed during informed consent
* Refusal to consider ART initiation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-06; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Adverse events | assessed at month 6 in each arm
  Any adverse events, such as confidentiality breaches, as a result of study participation

SECONDARY OUTCOMES:
MEMS adherence | assessed at months 3 and 6 in each arm
  Adherence to antiretroviral therapy, measured by MEMS Caps
plasma viral load | assessed at months 3 and 6 in each arm
  plasma HIV-1 RNA level

CONTACTS AND LOCATIONS:
Overall Officials: Susan M Graham, MD MPH PhD, Principal Investigator — University of Washington
Locations (1):
- Kenya Medical Research Institute Mtwapa Research Clinic, Mtwapa, Kenya

IPD SHARING:
Plan to Share IPD: Yes
Study data will be available after publication of the main study manuscripts. Researchers requesting access to data/resources will be asked to submit a request in writing describing their qualifications including their certification by their local IRB, analytic plans and other uses of the data/resources, and plans to secure the confidentiality and safety of the data. Given the sensitive nature of the data we are collecting, including HIV diagnosis and mental health status, we will not create a public access file.
Supporting Information: Study Protocol, ICF
Time Frame: Available from July 2017 for 2 years
Access Criteria: Researchers requesting access to data/resources will be asked to submit a request in writing describing their qualifications including their certification by their local IRB, analytic plans and other uses of the data/resources, and plans to secure the confidentiality and safety of the data.

REFERENCES:
- [Background] Graham SM, Micheni M, Kombo B, Van Der Elst EM, Mugo PM, Kivaya E, Aunon F, Kutner B, Sanders EJ, Simoni JM. Development and pilot testing of an intervention to promote care engagement and adherence among HIV-positive Kenyan MSM. AIDS. 2015 Dec;29 Suppl 3(0 3):S241-9. doi: 10.1097/QAD.0000000000000897. PMID 26562813